CLINICAL TRIAL: NCT00964561
Title: A Phase I, Single Blind, Randomized, Placebo Controlled, Drug Interaction Study of Intravenous (IV) Valortim® and Intravenous (IV) Ciprofloxacin in Healthy, Normal Subjects
Brief Title: Ph1 Study of Valortim and Ciprofloxacin in Humans
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: On partial hold for clinical investigation into AE and SAE reported.
Sponsor: PharmAthene, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); Medarex (Industry); Quintiles, Inc. (Industry); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Valerie Riddle, M.D., Vice President and Medical Director, PharmAthene, Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #0036-08-05; NIAID #08-0053
Record Dates: First submitted 2009-08-22; First posted 2009-08-25 (Estimated); Last update posted 2010-08-10 (Estimated); Status verified 2009-08

CONDITIONS: Anthrax
MeSH Terms: conditions — Anthrax | interventions — Ciprofloxacin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Ciprofloxacin and Valortim (Experimental): First two subjects to receive treatment arm of Ciprofloxacin and Valortim. Total of sixteen volunteers to be randomized to receive Ciprofloxacin and Valortim.
  Interventions: Drug: Ciprofloxacin and Valortim
- Placebo Antibiotic and Valortim (Experimental): Randomized such that four subjects to receive Placebo Antibiotic and Valortim.
  Interventions: Drug: Placebo Antibiotic and Valortim
- Placebo Antibiotic and Placebo Valortim (Experimental): Randomized such that 4 subjects to receive Placebo Antibiotic and Placebo Valortim.
  Interventions: Other: Placebo Antibiotic and Placebo Valortim

INTERVENTIONS:
Drug: Ciprofloxacin and Valortim — Days 1-3 400mg IV Ciprofloxacin BID over 60 minutes. Day 4 20mg/kg Valortim IV over 60 minutes.
  Other Names: MDX-1303
  Arms: Ciprofloxacin and Valortim
Drug: Placebo Antibiotic and Valortim — Days 1-3 20mg/kg IV Normal Saline BID over 60 minutes. Day 4 20mg/kg Valortim IV over 60 minutes.
  Other Names: MDX-1303
  Arms: Placebo Antibiotic and Valortim
Other: Placebo Antibiotic and Placebo Valortim — Days 1-3 200mL IV Normal Saline for Placebo Antibiotic over 60 minutes. Day 4 200mL IV Normal Saline for Placebo Valortim over 60 minutes.
  Other Names: Saline
  Arms: Placebo Antibiotic and Placebo Valortim

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of short-term dosing of IV ciprofloxacin when administered concomitantly with IV Valortim in healthy normal human subjects.

DETAILED DESCRIPTION:
Valortim (MDX-1303) is a fully human monoclonal antibody (hmAb) with a high affinity for B. anthracis protective antigen (PA). Valortim is designed to target PA, which is one of three plasmid-encoded proteins that together form the toxins released by B. anthracis. Individually, these proteins (protective antigen (PA), lethal factor (LF) and edema factor (EF)) are inactive. Toxic effects require the transport of LF and EF into the host cell, mediated by the activity of PA. Valortim binds to PA and interferes with the activity of the toxins. Based on both non-clinical and clinical data, Valortim may have utility for the pre- and post-exposure prophylaxis of individuals exposed to, or at risk of exposure to, B. anthracis and for the treatment of individuals displaying signs or symptoms of inhalational anthrax. Because the treatment of inhalational anthrax includes the use of antibiotics such as fluoroquinolones, it is necessary to demonstrate that there are no adverse interactions between newer therapeutic interventions and these medications. The purpose of this study is to assess the safety and pharmacokinetics of ciprofloxacin (a commonly used fluoroquinolone for both treatment and post-exposure prophylaxis of anthrax) and Valortim following co-administration, as well as the safety and tolerability of these medications when administered concomitantly. These data are intended to support the use of Valortim as a treatment for inhalational anthrax.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Normal male or female subjects 18 to 59 years of age on Day -1 of the study
2. Subject must have read, understood, and provided written informed consent after the nature of the study has been fully explained and must be willing to comply with all study requirements and procedures
3. In the opinion of the Investigator, subjects should be in generally good health, based upon prestudy medical history, physical examination, ECG and laboratory tests
4. Laboratory screening values (i.e., hematology, clinical chemistries and urinalysis tests) must be within study-defined ranges
5. No detectable antibody to B. anthracis Protective Antigen (PA-IgG) as measured by ELISA testing at study Screening
6. Women of childbearing potential may be enrolled if one of the following criteria applies:

   1. Must be using an effective form of contraception (e.g., oral contraceptives, vaginal ring, IUD, injected or implanted hormonal contraception, double barrier method of condom and spermicide, diaphragm with spermicide or sponge with spermicide) for at least one month prior to study entry, must have maintained a normal menstrual pattern for the three months prior to study entry and have a negative pregnancy test at the time of admission to the unit. Women must be willing to continue this contraception throughout the course of the study.
   2. Is sexually abstinent
   3. Is monogamous with a vasectomized partner (> 3 months prior)
   4. Is postmenopausal (i.e., no cycle for at least the previous 12 months, is of menopausal age (> 45 years) and has a negative urine pregnancy test prior to enrollment into the study and a negative serum pregnancy test on Day -1)
   5. Is surgically sterilized (confirmed by medical record review)
   6. Has had a total hysterectomy a minimum of 3 months prior to dosing on Day 1 (confirmed by medical record review)
7. Sexually active male subjects may be enrolled if one of the following criteria applies:

   1. Has had a vasectomy (> 3 months prior to study entry, confirmed by medical record review)
   2. Using condoms and whose partner is using an acceptable form of contraception (IUD, oral contraceptives, birth control patch or vaginal ring, injectable or implanted contraceptives, or tubal ligation [surgical sterilization]) for the duration of the study
   3. Is sexually abstinent
8. Female subjects must have a negative urine pregnancy test at study Screening and a negative serum pregnancy test on admission to the Phase I unit at Day -1
9. Female subject who are using injectable, transdermal, vaginal ring, oral contraceptives, or an IUD must agree to also use a barrier method (i.e. male condom, female condom, diaphragm, cervical cap) for the duration of their participation in the study.
10. Agreement to not receive any vaccinations from Day -1 through to 31 days post Valortim dosing. Vaccination against B. anthracis is prohibited during the study
11. Body Mass Index (BMI) ≥ 19 and ≤ 30
12. Abstinence from alcohol for 24 hours prior to study drug administration until discharge from the Phase I unit

Exclusion Criteria:

1. Prior known or suspected exposure to B. anthracis
2. Prior vaccination for B. anthracis
3. Any participants in the original FTIH study of Valortim.
4. History of drug or alcohol abuse i.e. having been treated either in an in-patient or out-patient facility within 12 months of study Screening
5. Positive drug result and/or positive alcohol result at time of study Screening or at Day -1
6. Smoke more than 10 cigarettes per day for the last 6 months
7. Treatment with an investigational agent within 30 days or 5 half-lives (whichever is longer) of study Screening
8. Use of systemic immunosuppressive agents within 12 months of study Screening. Individuals who have received prednisone or its equivalent in doses of less than 20 mg/day for 14 days or less, as long as it occurred more than 1 month prior to them entering the study and as long as there is no clinical or laboratory evidence of immunosuppression, may be considered for enrollment
9. Use of NSAIDs within 24 hours prior to dosing
10. History of asthma requiring any use of inhaled or oral medication within the previous 5 years
11. History of renal impairment
12. History of central nervous system reactivity to any quinolone
13. Any factor known to increase the risk of tendinitis or tendon rupture when taking a fluoroquinolone, including age older than 59 years; organ transplantation; use of systemic steroids (see number 7)
14. Clinically significant medical or psychiatric condition that, in the opinion of the Investigator, may impair study participation to include ongoing recent illness, new medications prescribed in the previous 6 weeks or use of immunosuppressive agents
15. Electrocardiogram with evidence of clinically significant conduction abnormalities or active ischemia (as determined by the Principal Investigator) at the time of study screening
16. Donation of one or more pints of blood 30 days prior to study Screening visit or donation prior to completion of Day 31 of the study
17. Donation of plasma within 14 days prior to study Screening visit or donation prior to completion of Day 31 of the study
18. Vaccinations within 30 days prior to Day -1 through to 31 days post Valortim dosing on Day 3
19. Prior known serum positivity for human immunodeficiency virus (HIV) antibodies, hepatitis B (surface antigen) or hepatitis C as determined at study Screening
20. Prior known allergy or allergic reaction to ciprofloxacin or any of the group of antibiotics known as quinolones
21. Diagnosis of photosensitivity, including, but not limited to, a history of phototoxic and/or photoallergic reactions to medications
22. Current treatment with, or use of, theophylline, methylxanthines, tizanidine, phenytoin, sulfonylurea glyburide, warfarin, probenecid, methotrexate, metoclopramide, corticosteroids and non-steroidal anti-inflammatory drugs
23. History of seizures, excluding pediatric febrile seizures

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2009-08; Primary Completion 2010-02 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Determination of changes from baseline for clinical laboratory tests and urinalysis, blood pressure, heart rate, respiratory rate, body temperature, physical examination and ECG | 134 days

SECONDARY OUTCOMES:
Evaluation of PK parameters for IV administration of ciprofloxacin when dosed concomitantly with Valortim | 134 days

CONTACTS AND LOCATIONS:
Overall Officials: Ralph A. Schutz, M.D., Principal Investigator — Quintiles, Inc.
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States

REFERENCES:
- See also: Go to this website for more information about this study. — http://www.studyforchange.com